CLINICAL TRIAL: NCT01197833
Title: A Multicenter, Randomized, Blinded Study of Endovenous Thermal Ablation With or Without Varisolve™ Polidocanol Endovenous Microfoam (PEM) Treatment for Patients With Great Saphenous Vein Incompetence and Visible Varicosities
Brief Title: Endovenous Ablation With and Without Polidocanol Endovenous Microfoam Treatment for Patients With Great Saphenous Vein Incompetence and Visible Varicosities
Acronym: 017
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAP.VV017
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Great Saphenous Vein Incompetence; Visible Varicosities
Keywords: varicose veins; Great saphenous vein; varicosities
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Endovenous ablation+polidocanol injectable microfoam 0.125% (Experimental): Endovenous ablation followed by an injection of polidocanol injectable microfoam 0.125% to target vein
  Interventions: Drug: endovenous ablation+polidocanol injectable microfoam 0.125%
- Endovenous ablation+polidocanol injectable micrfoam, 1.0% (Experimental): Endovenous ablation followed by injection of polidocanol injectable microfoam, 1.0% to the target vein
  Interventions: Drug: Endovenous ablation+polidocanol injectable microfoam 1.0%
- endovenous ablation+vehicle (placebo) (Active Comparator): endovenous ablation followed by injection of vehicle (placebo) to target vein
  Interventions: Drug: Endovenous ablation+polidocanol injectable foam 2.0%

INTERVENTIONS:
Drug: endovenous ablation+polidocanol injectable microfoam 0.125% — All components except API
  Other Names: endovenous ablation followed by polidocanol endovenous microfoam 0.125% injection to target vein
  Arms: Endovenous ablation+polidocanol injectable microfoam 0.125%
Drug: Endovenous ablation+polidocanol injectable microfoam 1.0% — endovenous ablation to target vein, followed by injection of polidocanol injectable foam 1.0%
  Other Names: Endovenous ablation followed by injection of polidocanol injectable foam 1.0% to target vein
  Arms: Endovenous ablation+polidocanol injectable micrfoam, 1.0%
Drug: Endovenous ablation+polidocanol injectable foam 2.0% — Endovenous ablation to target vein followed by injection of polidocanol injectable foam 2.0%
  Other Names: Endovenous ablation to target vein followed by injection of polidocanol injectable foam 2.0%
  Arms: endovenous ablation+vehicle (placebo)

SUMMARY:
Varicose veins are enlarged, noticeably bulging veins, which commonly occur in the legs and may cause discomfort. In this study, patients with varicose veins in the legs will be participating. The purpose of this research study is to evaluate the safety and effectiveness of two different doses of an investigational drug, Polidocanol Endovenous Microfoam (PEM) compared to vehicle (inactive solution) when used following an approved heat treatment in subjects with varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Incompetence of SFJ
* Patients who are candidates for ETA [laser or radiofrequency ablation (RFA)]
* Symptomatic varicose veins
* Visible varicose veins
* Ability to comprehend and sign an informed consent and complete study questionnaires in English

Exclusion Criteria:

* Patients who only have telangiectatic or reticular veins (Clinical Finding C1, as assessed by CEAP Classification of Venous Disorders)
* Patients who have active ulceration on the leg to be treated (Clinical Finding C6, as assessed by CEAP Classification of Venous Disorders)
* Leg obesity impairing the ability to access the vein to be treated and/or to apply post-procedure compression bandaging and stockings
* Ultrasonographic or other evidence of current or previous deep vein thrombosis or occlusion
* Deep venous reflux unless clinically insignificant in comparison to superficial reflux
* Peripheral arterial disease precluding the wearing of post-procedure compression bandaging and stockings
* Reduced mobility
* History of deep vein thrombosis, pulmonary embolism or stroke, including evidence of prior DVT on duplex ultrasound
* Major surgery, prolonged hospitalization or pregnancy within 3 months of screening
* Major co-existing disease (e.g. malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.)
* Known allergic response to polidocanol or heparin, including history of heparin-induced thrombocytopenia, and/or multiple allergic reactions
* Current alcohol or drug abuse
* Pregnant or lactating women
* Women of childbearing potential not using effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Scottsdale, Arizona
  - Bradenton, Florida
  - Oak Brook, Illinois
  - North Tonawanda, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Kirkland, Washington

REFERENCES:
- [Derived] Vasquez M, Gasparis AP; Varithena(R) 017 Investigator Group. A multicenter, randomized, placebo-controlled trial of endovenous thermal ablation with or without polidocanol endovenous microfoam treatment in patients with great saphenous vein incompetence and visible varicosities. Phlebology. 2017 May;32(4):272-281. doi: 10.1177/0268355516637300. Epub 2016 Mar 7. PMID 26957489

RESULTS

PARTICIPANT FLOW:
Groups:
- Endovenous Ablation, Vehicle Placebo: Endovenous ablation followed by vehicle placebo
- Endovenous Ablation, Polidocanol Injectable Foam, 0.5%: Endovenous ablation followed by polidocanol injectable foam, 0.5%
- Endovenous Ablation, Polidocanol Injectable Foam 1.0%: endovenous ablation followed by polidocanol injectable foam 1.0%
Period: Overall Study
Arm/Group | Endovenous Ablation, Vehicle Placebo | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% | Endovenous Ablation, Polidocanol Injectable Foam 1.0%
Started | 38 | 39 | 40
Completed | 38 | 39 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: all treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Endovenous Ablation, Vehicle Placebo | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% | Endovenous Ablation, Polidocanol Injectable Foam 1.0% | Total
Number analyzed (Participants) | 38 | 39 | 40 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.05) | 50.1 (11.60) | 51.8 (9.75) | 52.0 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 26 | 81
  Male | 12 | 10 | 14 | 36
BMI [Mean (Standard Deviation); unit: kg^m2] | 29.3 (6.04) | 27.7 (4.58) | 28.1 (5.25) | 28.3 (5.32)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Independent Photography Review (IPR-V3 Score)
Description: The Independent Photography Review - Visible Varicose Veins (IPR-V3) instrument is a 5-point scale used to assess the appearance of a patient's visible varicose veins. At screening, the site clinician was instructed to review the appearance of the patient's varicose veins in the medial section of each leg (a 'live' assessment), then select an IPR-V3 score (i.e., none=0, mild, moderate, severe or very severe=4) that best represented the appearance of the patient's varicose veins. This assessment took into account the attributes caliber, dilatation, tortuosity, and extent and number of varicosities, and was used to determine patient eligibility. The site clinician used a set of reference photographs (2 example photographs for each score on the scale) to assist with assigning a score to the appearance of the patient's visible varicose veins.
Time Frame: IPR-V3 measured at baseline and then at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Endovenous Ablation, Vehicle Placebo | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% | Endovenous Ablation, Polidocanol Injectable Foam 1.0%
Number analyzed (Participants) | 38 | 39 | 40
score | -0.80 (0.102) | -1.30 (0.100) | -1.11 (0.097)

2. Primary Outcome: Absolute Change From Baseline in PA-V3 Score
Description: The Patient Self-assessment of Visible Varicose Veins (PA-V3) instrument is a 5-point scale used by patients to evaluate the appearance of their visible varicose veins. On this paper questionnaire, the instructions included a diagram of the medial view of a leg with the area between the ankle and the groin circled. The patient was instructed to choose 1 of 5 response options that best described the appearance of the visible varicose veins of the leg that was treated in the study. The patient was instructed not to consider the appearance of the leg outside the circled area or of any spider veins. Possible responses ranged from "Not at all noticeable" (a score of 0) to "Extremely noticeable" (a score of 4)
Time Frame: PA-V3 measured at baseline and then at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Endovenous Ablation, Vehicle Placebo | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% | Endovenous Ablation, Polidocanol Injectable Foam 1.0%
Number analyzed (Participants) | 38 | 39 | 40
score | -1.59 (0.142) | -1.81 (0.140) | -1.85 (0.136)

ADVERSE EVENTS:
Arm/Group | Endovenous Ablation, Vehicle Placebo | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% | Endovenous Ablation, Polidocanol Injectable Foam 1.0%
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 20/38 | 29/39 | 35/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovenous Ablation, Vehicle Placebo (N=38) | Endovenous Ablation, Polidocanol Injectable Foam, 0.5% (N=39) | Endovenous Ablation, Polidocanol Injectable Foam 1.0% (N=40)
extravasation (General disorders) | 1 (1) | 3 (3) | 2 (2)
infusion site thrombosis (General disorders) | 0 (0) | 3 (3) | 3 (3)
edema peripheral (General disorders) | 0 (0) | 1 (1) | 4 (4)
tenderness (General disorders) | 0 (0) | 0 (0) | 3 (3)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 5 (5)
excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
pain in extermity (Musculoskeletal and connective tissue disorders) | 11 (11) | 14 (14) | 11 (11)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4)
deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
thrombophlebitis superficial (Vascular disorders) | 0 (0) | 13 (13) | 15 (15)
thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No